CLINICAL TRIAL: NCT05385601
Title: Eye Movements Recording Using a Smartphone: Comparison to Standard Video-oculography and Correlation to Imaging Data in Young Athletes
Status: Completed | Type: Observational
Sponsor: Association de Recherche Bibliographique pour les Neurosciences (Other)
Collaborators: Centre Hospitalier Princesse Grace (Other); Centre Hospitalier Universitaire de Nice (Other); Association Sportive Monaco Football Club (Unknown)
Responsible Party: Sponsor
Other Study IDs: e-VOG-Young Athletes-Extension
Record Dates: First submitted 2022-05-18; First posted 2022-05-23 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Healthy
Keywords: Young athletes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy young athletes (Eye-Tracker®T2 + e-VOG): Subjects who first perform standard video-oculography assessment, followed by e-VOG digital assessment.
  Interventions: Other: eVOG (Mobile VideoOculoGraphy)
- Healthy young athletes (e-VOG + Eye-Tracker®T2): Subjects who first perform e-VOG digital assessment, followed by the standard video-oculography assessment.
  Interventions: Other: eVOG (Mobile VideoOculoGraphy)

INTERVENTIONS:
Other: eVOG (Mobile VideoOculoGraphy) — * Eyes movements assessed with e-VOG (mobile application developed on an iPad, that uses the face detection features of the front camera to detect and record eye movements).
  * Study duration is about 20 minutes, the day the subject performs his standard video-oculography examination in routine care (using Eye-Tracker®T2)

SUMMARY:
This study aims to compare measurements obtained through the e-VOG application (mobile application, usable on smartphones or tablets, to record eye movements) with measurements from the standard video-oculography device (Eye-Tracker®T2), in young athletes. This study also aims to correlate these measurements with volumetric data from cerebral imaging (if MRI done in routine care at the same period, more or less 1 month).

DETAILED DESCRIPTION:
e-VOG Young athletes is a collaborative study between the Memory Center of the Rainier III Center (Princess Grace Hospital, Monaco), the Neurology Department of Nice University Hospital (France), and the AS Monaco Football Academy medical team.

Memory Center of the Rainier III Center is expert in eye-tracking and is equipped with a standard video-oculography device (Eye-Tracker®T2), which records eye movements at a high frequency and measures saccades parameters (latency, speed, amplitudes etc...).

e-VOG is a mobile application, home-developed by the Neurology Department team of Nice University Hospital, to measure eye movements.

In the continuity of the e-VOG(YA) study (NCT05211752), we set-up study named e-VOG-Young Athletes-Extension. This study will increase the number of assessments carried out (standard video-oculography assessment versus e-VOG digital assessment) in a population of athletes without major health problems, and who have not presented concussion, in order to meet more powerfully the main objective of the e-VOG(YA) study. It will also make it possible to observe whether there is a correlation between disturbed oculomotor movements, oculomotor anomalies and volumetric data measured by cerebral MRI (obtained using automatic segmentation software on cerebral regions specifically involved in the eye movement control).

ELIGIBILITY:
Inclusion Criteria:

* Young Athletes from AS Monaco Academy
* referred by AS Monaco Medical Team to perform a video-oculography (Eye-Tracking) examination as part of routine care.
* covered by a health insurance system
* volunteer, able to give free, informed and written consent.

Exclusion Criteria:

* General anaesthesia within 3 months.
* Head trauma within 3 months
* Neurological, ophthalmological or general pathology preventing the realization of a video-oculography examination.
* Oculomotor abnormality detectable on clinical examination by the neurologist prescribing the standard video-oculography examination.

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Young athletes for whom a standard video-oculography exam is prescribed by the AS Monaco Football medical Team as part of a preventive and follow-up approach performed in routine care.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-06-08 (Actual)

PRIMARY OUTCOMES:
Oculomotor profiles concordance | Day 0
  Analyze of the concordance of the profiles obtained between the e-VOG digital assessment and the standard video-oculography assessment.
  Evaluation criteria: For each assessment, patients will be classified according to the number of oculomotor abnormality observed (based on identified parameters assessments: latency / speed / gain / altered ocular pursuits / fixation disorders / presence of internuclear ophthalmoplegia), in accordance with the literature standards

SECONDARY OUTCOMES:
Latency during horizontal reflex saccades | Day 0
  Measure of Latency during an horizontal reflex saccades paradigm with e-VOG Compared to the one performed with standard video-oculography device.
  Evaluation criteria: latency (reaction time in ms).
Latency during vertical reflex saccades | Day 0
  Measure of Latency during a vertical reflex saccades paradigm with e-VOG Compared to the one performed with standard video-oculography device.
  Evaluation criteria: latency (reaction time in ms).
Latency during horizontal voluntary saccades | Day 0
  Measure of Latency during an horizontal volontary saccades paradigm with e-VOG Compared to the one performed with standard video-oculography device.
  Evaluation criteria: latency (reaction time in ms).
Velocity during horizontal reflex saccades | Day 0
  Measure of Velocity during an horizontal reflex saccades paradigm with e-VOG Compared to the one performed with standard video-oculography device.
  Evaluation criteria: velocity (mean and peak velocity) in °/s.
Velocity during vertical reflex saccades | Day 0
  Measure of Velocity during a vertical reflex saccades paradigm with e-VOG Compared to the one performed with standard video-oculography device.
  Evaluation criteria: velocity (mean and peak velocity) in °/s.
Inhibition capacity | Day 0
  Measure of inhibition capacity performance during an antisaccades" paradigm with e-VOG Compared to the one evaluated with standard video-oculography device.
  Evaluation criteria: percentage of errors.
Internuclear ophthalmoplegia (INO) detection | Day 0
  Highlight presence/absence of INO with e-VOG Compared to standard video-oculography device.
  Evaluation criteria: INO is present if calculated ratio of abducting to adducting eye movement (both mean and peak velocity) is >1.
Fixations impairments detection | Day 0
  Highlight presence/absence of Fixations impairments with e-VOG Compared to standard video-oculography device.
  Evaluation criteria: presence/absence/frequency of square wave-jerks, nystagmus, flutters.
Impairment of horizontal smooth pursuit | Day 0
  Highlight Impairment of horizontal smooth pursuit with e-VOG Compared to standard video-oculography device.
  Evaluation criteria: presence/absence of saccade and perturbation.
Impairment of vertical smooth pursuit | Day 0
  Highlight Impairment of horizontal smooth pursuit with e-VOG Compared to standard video-oculography device.
  Evaluation criteria: presence/absence of saccade and perturbation.
Imaging data correlation: Total brain volume | Day 0
  Analyze if there are correlation between oculomotor abnormalities and volumetric data measured by brain MRI.
  Evaluation criteria: Total brain volume (Data from cerebellar MRI performed in routine care, obtained using automatic segmentation software).
Imaging data correlation: Frontal Lobe Volume | Day 0
  Analyze if there are correlation between oculomotor abnormalities and volumetric data measured by brain MRI.
  Evaluation criteria: Frontal Lobe Volume (Data from cerebellar MRI performed in routine care, obtained using automatic segmentation software).
Imaging data correlation: Parietal Lobe Volume | Day 0
  Analyze if there are correlation between oculomotor abnormalities and volumetric data measured by brain MRI.
  Evaluation criteria: Parietal Lobe Volume (Data from cerebellar MRI performed in routine care, obtained using automatic segmentation software).
Imaging data correlation: Volume of additional motor areas | Day 0
  Analyze if there are correlation between oculomotor abnormalities and volumetric data measured by brain MRI.
  Evaluation criteria: Volume of additional motor areas (Data from cerebellar MRI performed in routine care, obtained using automatic segmentation software).
Imaging data correlation: Basal ganglia volume | Day 0
  Analyze if there are correlation between oculomotor abnormalities and volumetric data measured by brain MRI.
  Evaluation criteria: Basal ganglia volume (Data from cerebellar MRI performed in routine care, obtained using automatic segmentation software).
Imaging data correlation: Total thalamic volume | Day 0
  Analyze if there are correlation between oculomotor abnormalities and volumetric data measured by brain MRI.
  Evaluation criteria: Total thalamic volume (Data from cerebellar MRI performed in routine care, obtained using automatic segmentation software).
Imaging data correlation: cerebellar volume | Day 0
  Analyze if there are correlation between oculomotor abnormalities and volumetric data measured by brain MRI.
  Evaluation criteria: Cerebellar volume (Data from cerebellar MRI performed in routine care, obtained using automatic segmentation software).

CONTACTS AND LOCATIONS:
Overall Officials: Mikael COHEN, MD, Principal Investigator — Centre de Ressources et de Compétences SEP, UMRC Pasteur 2, Université Nice Côte d'Azur, Nice-France; Sandrine LOUCHART DE LA CHAPELLE, MD-PHD, Principal Investigator — Centre Mémoire, Centre de Gérontologie Clinique RAINIER III, Princess Grace Hospital, Monaco; Alain PESCE, MD-PHD, Study Director — AREBISN (Association de Recherche Bibliographique pour les Neurosciences), Nice (France)
Locations (1):
- Centre Mémoire / Centre de Gérontologie Clinique Rainier III / Princess Grace Hospital, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: No